CLINICAL TRIAL: NCT05758597
Title: Clinical Study on Sedative Effect and Safety of Remimazolam Besylate in ARDS Patients With Mechanical Ventilation
Brief Title: Sedative Effect and Safety of Remimazolam Besylate in ARDS Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhiming Jiang (Other)
Responsible Party: Sponsor-Investigator, Zhiming Jiang, Head of Critical Care Medicine, Qianfoshan Hospital of Shandong Province, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YXLL-KY-2022(105)
Record Dates: First submitted 2022-11-25; First posted 2023-03-07 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remazolam besylate group (Experimental): The remimazolam besylate treatment group was given remimazolam besylate 0.1-1mg/kg/h to maintain the target RASS score.
  Interventions: Drug: Remazolam besylate
- Midazolam group (Active Comparator): The midazolam treatment group was given midazolam 0.05-0.2 mg/kg/h to maintain the target RASS score.
  Interventions: Drug: midazolam

INTERVENTIONS:
Drug: Remazolam besylate — Remazolam benzoate group was given 0.1-1mg/kg/h, and the target RASS score was maintained.
  Other Names: Yichang Humanwell
  Arms: Remazolam besylate group
Drug: midazolam — Meanwhile the midazolam group was given 0.05-0.2 mg/kg/h midazolam, and the target RASS score was maintained.
  Other Names: Jiangsu ehwa
  Arms: Midazolam group

SUMMARY:
The incidence and mortality of acute respiratory distress syndrome (ARDS) are high. Patients with ARDS often need mechanical ventilation. Rational use of sedation and analgesia can improve the tolerance of patients with mechanical ventilation and reduce the lung injury caused by mechanical ventilation. Currently, the main sedative drugs used in clinical practice are midazolam, propofol and dexmedetomidine, but they all have disadvantages. It is urgent to find a sedative drug that can achieve rapid and sufficient sedation, does not inhibit breathing, leads to rapid recovery after drug withdrawal and does not increase incidence of delirium.

Remimazolam besylate is a newly marketed ultra-short-acting GABAa receptor agonist, which is not metabolized by liver or kidney and is easily hydrolyzed by non-specific esterase in vivo. It has rapid effect, short recovery time, continuous infusion with almost no accumulation, little influence on respiration and circulation, and can be antagonized by flumasini. Compared with the above traditional sedatives, it has obvious advantages, especially suitable for sedation in ICU patients. There are few studies on remimazolam besylate used for sedation in ICU patients. At present, there is a lack of evidence-based medical evidence for the application of remazolam besylate in ICU patients. Its efficacy and safety, potential advantages and dominant population, application dose and combination of drugs still need to be further explored and clarified. The objective of this study was to investigate the sedative effects and advantages of remimazolam besylate versus midazolam in patients with ARDS requiring invasive mechanical ventilation. The successful undergoing of this study will provide practical basis for clinical sedation in patients with ARDS mechanical ventilation.

DETAILED DESCRIPTION:
The incidence and mortality of acute respiratory distress syndrome (ARDS) are high. Patients with ARDS often need mechanical ventilation. Rational use of sedation and analgesia can improve the tolerance of patients with mechanical ventilation and reduce the lung injury caused by mechanical ventilation. Currently, the main sedative drugs used in clinical practice are midazolam, propofol and dexmedetomidine, but they all have disadvantages. It is urgent to find a sedative drug that can achieve rapid and sufficient sedation, does not inhibit breathing, leads to rapid recovery after drug withdrawal and does not increase incidence of delirium. Remimazolam besylate is a newly marketed ultra-short-acting GABAa receptor agonist, which is not metabolized by liver or kidney and is easily hydrolyzed by non-specific esterase in vivo. It has rapid effect, short recovery time, continuous infusion with almost no accumulation, little influence on respiration and circulation, and can be antagonized by flumasini. Compared with the above traditional sedatives, it has obvious advantages, especially suitable for sedation in ICU patients. There are few studies on remimazolam besylate used for sedation in ICU patients. At present, there is a lack of evidence-based medical evidence for the application of remimazolam besylate in ICU patients. Its efficacy and safety, potential advantages and dominant population, application dose and combination of drugs still need to be further explored and clarified. The objective of this study was to investigate the sedative effects and advantages of remimazolam besylate versus midazolam in patients with ARDS requiring invasive mechanical ventilation. The successful undergoing of this study will provide practical basis for clinical sedation in patients with ARDS mechanical ventilation. Detailed Description: Reasonable and appropriate analgesic sedation can effectively reduce the incidence of anxiety, agitation and delirium in ICU patients, shorten length of mechanical ventilation and ICU stay, and improve the prognosis. Acute respiratory distress syndrome (ARDS) is a clinical syndrome caused by acute diffuse inflammatory injury of lung, which is induced by infection, shock, trauma, etc. Acute respiratory distress syndrome (ARDS) is present in 10% of patients admitted to the intensive care unit (ICU) and is associated with 35% to 46% of ICU in-patient mortality. Patients with ARDS need careful supportive treatment, including rational use of sedation and analgesia. Sedation and analgesia are beneficial to ARDS patients to some extent, which can improve the tolerance of mechanical ventilation, reduce oxygen consumption, and reduce lung injury caused by mechanical ventilation. The 2018 Chinese Guidelines for Analgesia and Sedation suggest that patients in the acute stage of stress with unstable organ functions should be given deeper sedation to protect organ functions. However, ventilator parameters (such as pressure control mode, retention of spontaneous breathing, reduced sensitivity to inspiratory triggers, etc.) should be adjusted prior to the formulation of sedation and analgesia to avoid the use of unnecessary deep sedation or neuromuscular blockers. At present, midazolam, propofol and dexmedetomidine are the main sedative drugs used in clinical practice. Midazolam has the characteristics of antianxiety and high rate of anterograde amnesia during sedation. Compared with other sedatives, prolonged mechanical ventilation is regarded as a risk factor for delirium in ICU patients. Propofol has been reported that after long-term infusion, its active metabolites are easy to accumulate in the body, which may lead to propofol infusion syndrome in severe cases . The sedative advantage of dexmedetomidine lies in that a large dose of dexmedetomidine does not inhibit respiratory drive, can achieve conscious sedation, and has a lower risk of delirium than midazolam. However, the use of dexmedetomidine cannot quickly achieve full sedation of patients, and the maximum dose of infusion recommended by the instructions is difficult to make the RASS score of patients lower than -3 , and may lead to decreased heart rate and blood pressure, which may affect tissue perfusion and other deficiencies . Therefore, there is an urgent need for a sedative agent that can achieve rapid and sufficient sedation, without inhibiting respiration, and allow patients to wake up quickly after drug withdrawal without increasing the patient's delirium. Ramimazolam besylate is an ultra-short-acting GABAa receptor agonist by acting on GABAa receptors, opening chloride ion channels to promote the internal flow of chloride ions, causing hyperpolarization of nerve cell membranes and inhibition of neurons. It can cause a decrease in body activity, sedation, amnesia and other effects. Remimazolam does not undergo liver or kidney metabolism and is easily hydrolyzed by non-specific esterase in vivo. It has the advantages of rapid onset, short recovery time, almost no accumulation of continuous infusion, little influence on respiration and circulation, and can be antagonized by flumasini. Compared with the above traditional sedative drugs, it is especially suitable for sedation in ICU patients. There are few studies on remimazolam besylate used for sedation in ICU patients. A clinical study on sedation of patients with mechanical ventilation in ICU showed that compared with propofol, Remimazolam besylate is more suitable for sedation of ICU patients because it has faster recovery and less impact on heart rate, blood pressure and cardiac systolic function. Goudra BG et al. proposed remimazolam besylate as the first choice for ICU sedation based on a large number of literature studies and analysis, which has great potential in the future. However, the use of remimazolam besylate in ICU patients is still lacking evidence-based medical evidence, and its efficacy and safety, potential advantages and advantaged population, dosage and combination of drugs still need to be further explored and clarified. The purpose of this study was to investigate the sedative effects and advantages of remimazolam besylate and the traditional sedative midazolam in patients with ARDS requiring invasive mechanical ventilation, in order to provide a practical basis for clinical sedation in patients with ARDS invasive mechanical ventilation. The secondary objective was to determine the incidence of associated adverse reactions and the changes of related biomarkers during sedation with remimazolam besylate in mechanical ventilation patients with ARDS This is a single-center, randomized, controlled prospective clinical study. It is expected that 100 patients will be enrolled, and 50 patients in each group will be randomly assigned by the network at a ratio of 1:1. Drugs were injected intravenously in both groups, the analgesic target CPOT score was less than 3 points, and the sedation target was set according to the respiratory mechanical goal: RASS score of the shallow sedation group was 0 ~ -2 points; Deep sedation group: RASS score -3 ~ -5 points. Remifentanil was given to maintain a CPOT score of less than 3 points. They were divided into remimazolam besylate group and midazolam group. Before medication, 30min, 4h, 8h, 12h, 24h, 48h after medication until the end point of visit (after drug withdrawal). The main study indicators are proportion of patients who achieved the target sedation level during the study observation time node, hemodynamic indexes, mechanical ventilation time, ICU stay time, mortality within 28 days at each observation time point, etc. The incidence of adverse reactions in the two groups was also assessed. Te stopping criteria included extubation, discharge from our ICU, discontinuation of study drugs for 24 h by treating physicians and 7 days after enrollment, whichever came frst. Patients were followed up for 28 days.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥18 years old and ≤65 years old
2. ARDS patients admitted to ICU requiring invasive mechanical ventilation (meeting the 2012 Berlin diagnostic criteria for ARDS)
3. Expected mechanical ventilation time > 3 days
4. Obtain informed consent from patients or family members

Exclusion Criteria:

1. Pregnancy or lactation
2. Patients with myasthenia gravis, acute myocardial ischemia or severe arrhythmia
3. Severe, pre-existing substantive liver disease with clinically significant portal hypertension, Child-Pugh C cirrhosis, or acute liver failure
4. Severe craniocerebral injury, brain tumor, increased intracranial pressure, cerebrovascular accident, coma, epilepsy, etc.
5. Patients with a history of alcohol or drug abuse or chronic pain requiring long- term use of analgesic and sedative drugs
6. Any conditions that interfere with the correct assessment of cognitive function, such as language and sensory disorders or mental disorders (language difficulties or organic mental dysfunction
7. Participate in other exploratory clinical trials within 3 months prior to screening
8. Known or suspected allergies to remazolam besylate, midazolam, propofol, and opioids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-16 (Estimated)

PRIMARY OUTCOMES:
Comparison of sedative effect | From the date of using of remimazolam besylate Until the date of extubation, discharge from our ICU, discontinuation of study drugs for 24 hours by treating physicians, whichever came frst，assessed up to 7 days
  Percentage of patients who achieved the target sedation range in different treatment groups
Comparison of respiratory status | Before medication
  Oxygenation index (PaO2/FiO2) in millimeters of mercury before medication
Comparison of respiratory status | 24 hours after medication
  Oxygenation index (PaO2/FiO2) in millimeters of mercury 24 hours after medication
Comparison of respiratory status | 48 hours after medication
  Oxygenation index (PaO2/FiO2) in millimeters of mercury 48 hours after medication
Comparison of length of stay in ICU | From the beginning of the study to transfer out of the ICU，assessed up to 30 days
  length of stay in ICU between different treatment groups
comparison of mortality | From the beginning of the study to the end of follow-up, assessed up to 3 months
  mortality in different treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Jiang, doctor, Study Director — Department of Intensive Care Medicine, Qianfoshan Hospital, Shandong Province
Locations (1):
- Department of Intensive Care Medicine, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Payen JF, Chanques G, Mantz J, Hercule C, Auriant I, Leguillou JL, Binhas M, Genty C, Rolland C, Bosson JL. Current practices in sedation and analgesia for mechanically ventilated critically ill patients: a prospective multicenter patient-based study. Anesthesiology. 2007 Apr;106(4):687-95; quiz 891-2. doi: 10.1097/01.anes.0000264747.09017.da. PMID 17413906
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Tan JA, Ho KM. Use of dexmedetomidine as a sedative and analgesic agent in critically ill adult patients: a meta-analysis. Intensive Care Med. 2010 Jun;36(6):926-39. doi: 10.1007/s00134-010-1877-6. Epub 2010 Apr 8. PMID 20376429
- [Background] Shehabi Y, Ruettimann U, Adamson H, Innes R, Ickeringill M. Dexmedetomidine infusion for more than 24 hours in critically ill patients: sedative and cardiovascular effects. Intensive Care Med. 2004 Dec;30(12):2188-96. doi: 10.1007/s00134-004-2417-z. Epub 2004 Aug 26. PMID 15338124
- [Background] Zhang Z, Chen K, Ni H, Zhang X, Fan H. Sedation of mechanically ventilated adults in intensive care unit: a network meta-analysis. Sci Rep. 2017 Mar 21;7:44979. doi: 10.1038/srep44979. PMID 28322337
- [Background] Goudra BG, Singh PM. Remimazolam: The future of its sedative potential. Saudi J Anaesth. 2014 Jul;8(3):388-91. doi: 10.4103/1658-354X.136627. PMID 25191193